CLINICAL TRIAL: NCT02003664
Title: A Randomized Placebo-controlled Study of Baclofen ER on Brain and Behavioral Outcomes in Cocaine Dependence
Brief Title: A Study of Baclofen ER
Acronym: CURE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study never started due to delays in medication development
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 819017
Record Dates: First submitted 2013-11-19; First posted 2013-12-06 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Treatment; fMRI; Outcomes
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen ER versus Placebo (Active Comparator): Baclofen ER versus Placebo (sugar pill)
  Interventions: Drug: Baclofen ER
- Placebo versus Baclofen ER (Placebo Comparator): Participants will receive either placebo (sugar pill) or Baclofen ER
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen ER — Comparison of Baclofen ER to placebo using a 2 to 1 chance of receiving Baclofen ER, the medication
  Arms: Baclofen ER versus Placebo
Drug: Placebo — Comparison of placebo to Baclofen ER using a 1 in 3 chance of receiving placebo
  Other Names: Sugar pill
  Arms: Placebo versus Baclofen ER

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled study that will examine the efficacy of extended-release baclofen (Baclofen ER) for the treatment of cocaine dependence. The primary study outcome will be urines positive for benzoylecgonine (BE), a metabolite of cocaine, submitted during outpatient treatment (12-week) and follow-up (12-week). To examine brain mechanisms of relapse/recovery, participants will complete fMRI sessions before, during, and after treatment. Brain responses to specific probes of reward and inhibition will be used as biomarkers predicting drug use during and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Physically healthy cocaine-dependent (based on DSM-IV- TR criteria) male or female aged 18-60 yrs, voluntarily seeking treatment for cocaine dependence.
2. Females must be non-pregnant, non- lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of child bearing potential, but practicing a medically acceptable method of birth control. Examples of medically acceptable methods for this protocol include barrier (diaphragm or condom) with spermicide, an intrauterine device (IUD), oral contraceptives, a levonorgestrel implant, intrauterine progesterone contraceptive system, medroxyprogesterone acetate contraceptive injection, and abstinence.
3. Reading level at or above eighth grade.
4. Participants provide voluntary informed consent.
5. Smoking is primary route of cocaine administration.
6. Available for an inpatient stay.

Exclusion Criteria:

1. Participation in clinical trial and receipt of investigational drug(s) during previous 60 days, except as explicitly approved by the Principal Investigator.
2. Clinically significant cardiovascular, hematologic, hepatic, renal, neurological or endocrinological abnormalities.
3. History of serious head trauma or injury causing loss of consciousness that lasted more than 3 minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI.
4. Presence of magnetically active prosthetics, plates, pins, broken needles, permanent retainer, bullets, etc. in patient's body (unless a radiologist confirms that its presence is unproblematic). An x-ray may be obtained to determine eligibility.
5. Claustrophobia or other medical condition that disables the participant from lying in the MRI for approximately 60 minutes.
6. Current or prior gambling problems (assessed by participants self-report)
7. Non-removable skin patches
8. Have received medication that could interact adversely with baclofen, including muscle relaxants (including tricyclic antidepressants), antiseizure medication, CNS depressants (tranquilizers, sleeping pills), MAO inhibitors), within the time of administration of study agent based on the study physician's guidance (e.g. 5 half lives)
9. Have known or suspected hypersensitivity to baclofen.
10. Be taking baclofen for any reason currently or during the past year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Urines positive for benzoylecgonine (BE), (a metabolite of cocaine) | up to 24 weeks
  The primary clinical outcome is number of cocaine-use days (assessed by urines positive for benzoylecgonine (BE), a metabolite of cocaine) during the outpatient treatment and follow-up phases of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rose Childress, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for the Studies of Addiction, Philadelphia, Pennsylvania, United States